CLINICAL TRIAL: NCT02994368
Title: A Multicenter Prospective Observational "Natural History" Study in Patients With Choroideremia
Brief Title: "Natural History" Study of Choroideremia
Status: Terminated | Type: Observational
Sponsor: 4D Molecular Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: 4D-CHM-001-NH-0001
Record Dates: First submitted 2016-12-13; First posted 2016-12-15 (Estimated); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Choroideremia
Keywords: retinal degeneration; eye; REP-1 gene
MeSH Terms: conditions — Choroideremia; Retinal Degeneration | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Primary Cohort: No intervention
  Interventions: Other: Observation
- Expansion Cohort: No intervention
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation

SUMMARY:
The purpose of this study is to understand the rate of progression of all stages of choroideremia using a variety of assessments performed in the clinic including visual field measures, specialized photography of the eye and participant-reported visual problems

ELIGIBILITY:
Inclusion Criteria (Primary Cohort):

* Healthy individuals (at least 14 years) with choroideremia (20/200 or better vision) willing to participate in an observational study and meeting the eligibility criteria.

Inclusion Criteria (Expansion Cohort):

* Healthy individuals (at least 18 years) with choroideremia (20/200 or better vision in both eyes) willing to participate in an observational study and meeting the eligibility criteria.

Exclusion Criteria (Primary and Expansion Cohort):

1. Prior therapy with an AAV vector-based treatment
2. Pre-existing eye conditions that would: (1) preclude future planned treatment in a therapeutic intent clinical trial (i.e. intravitreal injection), (2) interfere with the interpretation of study endpoints, and/ or put patient at risk for surgical complications
3. Complicating systemic diseases that would preclude future enrollment in a therapeutic intent clinical trial
4. Any other condition that would not allow the potential subject to complete follow-up examinations during the course of the study and, in the opinion of the investigator, makes the potential subject unsuitable for the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with a clinical diagnosis of choroideremia
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2016-12; Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Rate of progression of disease | 4 years
  A variety of psychophysical, anatomical and image-based endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Schonmei Lee, MD, Study Director — 4D Molecular Therapeutics
Locations (4):
- United States (3):
  - Retina Foundation of the Southwest, Dallas, Texas
  - Baylor College of Medicine, Ophthalmology-Cullen Eye Center, Houston, Texas
  - Moran Eye Center, University of Utah, Salt Lake City, Utah
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No